CLINICAL TRIAL: NCT05680675
Title: Dual-Tracer Theranostic PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: MultiFunctional Imaging LLC (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI158172; 2R44CA257522 (NIH)
Record Dates: First submitted 2022-12-22; First posted 2023-01-11 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Neuroendocrine Tumors; Prostate Cancer
Keywords: somatostatin receptor-positive
MeSH Terms: conditions — Neuroendocrine Tumors; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): Single-Tracer FDG (F18 Fluorodeoxyglucose) PET/CT exam + Single-Tracer Cu64-DOTATATE PET/CT
  Interventions: Diagnostic Test: Single-Tracer FDG PET/CT Exam; Diagnostic Test: Single-Tracer Cu64-DOTATATE PET/CT Exam
- Arm 2 (Experimental): Single-Tracer FDG PET/CT exam + Single-Tracer Ga68-DOTATATE PET/CT exam
  Interventions: Diagnostic Test: Single-Tracer FDG PET/CT Exam; Diagnostic Test: Single-Tracer Ga68-DOTATATE PET/CT Exam
- Arm 3 (Experimental): Single-Tracer FDG PET/CT exam + Single-Tracer PSMA (prostate-specific membrane antigen) PET/CT exam
  Interventions: Diagnostic Test: Single-Tracer FDG PET/CT Exam; Diagnostic Test: Single-Tracer PSMA PET/CT Exam

INTERVENTIONS:
Diagnostic Test: Single-Tracer FDG PET/CT Exam — The PET technologist will administer approximately 15 millicuries (mCi) of FDG intravenously, and the participant will remain resting during the tracer uptake period. A CT topogram will be obtained, and the PET imaging field-of-view (FOV) selected. The PET scan will then be acquired, acquiring 5 back-to-back "whole-body" (eyes-to-thighs, or similar) scans, providing 5 sequential PET images.
Diagnostic Test: Single-Tracer Cu64-DOTATATE PET/CT Exam — The PET technologist will administer with approximately 4 mCi Cu64-DOTATATE intravenously, and the participant will remain resting during the tracer uptake period. A CT topogram will be obtained, and the PET imaging field-of-view (FOV) selected. The PET scan will then be acquired, acquiring 5 back-to-back "whole-body" (eyes-to-thighs, or similar) scans, providing 5 sequential PET images.
  Arms: Arm 1
Diagnostic Test: Single-Tracer Ga68-DOTATATE PET/CT Exam — The PET technologist will administer with with approximately 5 mCi Ga68-DOTATATE intravenously, and the participant will remain resting during the tracer uptake period. A CT topogram will be obtained, and the PET imaging field-of-view (FOV) selected. The PET scan will then be acquired, acquiring 5 back-to-back "whole-body" (eyes-to-thighs, or similar) scans, providing 5 sequential PET images.
  Arms: Arm 2
Diagnostic Test: Single-Tracer PSMA PET/CT Exam — The PET technologist will administer with with approximately 7 mCi Ga68-PSMA-11 intravenously, and the participant will remain resting during the tracer uptake period. A CT topogram will be obtained, and the PET imaging field-of-view (FOV) selected. The PET scan will then be acquired, acquiring 5 back-to-back "whole-body" (eyes-to-thighs, or similar) scans, providing 5 sequential PET images.
  Arms: Arm 3

SUMMARY:
This study is designed to obtain positron emission tomography with x-ray computed tomography (PET/CT) imaging data with each tracer pair, providing the imaging data needed to develop new simultaneous dual-tracer imaging techniques and processing algorithms for these tracer pairs.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 years or greater.
* willing and able to sign a written informed consent and HIPAA authorization in accordance with local and institutional guidelines.
* presence of at least 1 measurable lesion ≥ 1 cm in size.
* willing to have their clinical records reviewed for at least 24 months after enrollment.
* willing to lie flat on their back in the PET/CT scanner for up to one hour to allow for the imaging data to be obtained.
* willing to undergo two separate PET/CT exams on different days within 2 weeks of each other.
* female participants who are not postmenopausal or surgically sterile will undergo a serum pregnancy test prior to baseline and the subsequent set of multi-tracer PET scans. The serum pregnancy test must be performed within 48 hours prior to research PET imaging. A negative test will be necessary for such patients to undergo research PET imaging. This only applies to Arms 1 and 2, since only males will be included in Arm 3 (only males can get prostate cancer).
* Arms 1 and 2 only: known or suspected somatostatin receptor-positive neuroendocrine tumor (NET) who could be considered for clinical use of DOTATATE PET/CT imaging under the approved indications for use of this radiopharmaceutical according to published appropriate use criteria. These indications include initial staging after the histologic diagnosis of NET, evaluation of an unknown primary; evaluation of a mass suggestive of NET not amenable to endoscopic or percutaneous biopsy, staging of NET before planned surgery, monitoring of NET seen predominantly on somatostatin receptor (SSTR) PET, evaluation of patients with biochemical evidence and symptoms of a NET, evaluation of patients with biochemical evidence of a NET without evidence on conventional imaging or a prior histologic diagnosis, restaging at time of clinical or laboratory progression without progression on conventional imaging, and new indeterminate lesion on conventional imaging with unclear progression.
* Arm 3 Only: known or suspected prostate cancer who could be considered for clinical use of PSMA PET/CT imaging under the approved indications for use of this radiopharmaceutical, including patients with suspected metastasis and patients with suspected recurrence based on elevated serum prostate-specific antigen (PSA) level.

Exclusion Criteria:

* received somatostatin receptor targeted therapy at any time prior to enrollment will be excluded from the study Arms involving DOTATATE (Arms 1-2).
* known intolerance or hypersensitivity to any somatostatin analogs will be excluded from the study Arms involving DOTATATE (Arms 1-2).
* participated in any therapeutic clinical study or received any investigational agent within the last 30 days.
* known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals
* require monitored anesthesia for PET/CT scanning.
* too claustrophobic to undergo PET/CT scanning.
* exceed the 450 lb. weight limit of the PET/CT scanner.
* pregnant or currently breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Yap, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single-Tracer FDG (F18 Fluorodeoxyglucose) PET/CT + Single-Tracer Cu64-DOTATATE PET/CT Exams: Single-Tracer FDG PET/CT Exam: The PET technologist will administer approximately 15 millicuries (mCi) of FDG intravenously, and the participant will remain resting during the tracer uptake period. A CT topogram will be obtained, and the PET imaging field-of-view (FOV) selected. The PET scan will then be acquired, acquiring 5 back-to-back "whole-body" (eyes-to-thighs, or similar) scans, providing 5 sequential PET images.
  Single-Tracer Cu64-DOTATATE PET/CT Exam: The PET technologist will administer with approximately 4 mCi Cu64-DOTATATE intravenously, and the participant will remain resting during the tracer uptake period. A CT topogram will be obtained, and the PET imaging field-of-view (FOV) selected. The PET scan will then be acquired, acquiring 5 back-to-back "whole-body" (eyes-to-thighs, or similar) scans, providing 5 sequential PET images.
- Single-Tracer FDG PET/CT + Single-Tracer Ga68-DOTATATE PET/CT Exams: Single-Tracer FDG PET/CT Exam: The PET technologist will administer approximately 15 millicuries (mCi) of FDG intravenously, and the participant will remain resting during the tracer uptake period. A CT topogram will be obtained, and the PET imaging field-of-view (FOV) selected. The PET scan will then be acquired, acquiring 5 back-to-back "whole-body" (eyes-to-thighs, or similar) scans, providing 5 sequential PET images.
  Single-Tracer Ga68-DOTATATE PET/CT Exam: The PET technologist will administer with with approximately 5 mCi Ga68-DOTATATE intravenously, and the participant will remain resting during the tracer uptake period. A CT topogram will be obtained, and the PET imaging field-of-view (FOV) selected. The PET scan will then be acquired, acquiring 5 back-to-back "whole-body" (eyes-to-thighs, or similar) scans, providing 5 sequential PET images.
- Single-Tracer FDG PET/CT + Single-Tracer PSMA (Prostate-specific Membrane Antigen) PET/CT Exams: Single-Tracer FDG PET/CT Exam: The PET technologist will administer approximately 15 millicuries (mCi) of FDG intravenously, and the participant will remain resting during the tracer uptake period. A CT topogram will be obtained, and the PET imaging field-of-view (FOV) selected. The PET scan will then be acquired, acquiring 5 back-to-back "whole-body" (eyes-to-thighs, or similar) scans, providing 5 sequential PET images.
  Single-Tracer PSMA PET/CT Exam: The PET technologist will administer with with approximately 7 mCi Ga68-PSMA-11 intravenously, and the participant will remain resting during the tracer uptake period. A CT topogram will be obtained, and the PET imaging field-of-view (FOV) selected. The PET scan will then be acquired, acquiring 5 back-to-back "whole-body" (eyes-to-thighs, or similar) scans, providing 5 sequential PET images.
Period: Overall Study
Arm/Group | Single-Tracer FDG (F18 Fluorodeoxyglucose) PET/CT + Single-Tracer Cu64-DOTATATE PET/CT Exams | Single-Tracer FDG PET/CT + Single-Tracer Ga68-DOTATATE PET/CT Exams | Single-Tracer FDG PET/CT + Single-Tracer PSMA (Prostate-specific Membrane Antigen) PET/CT Exams
Started | 15 | 15 | 20
Completed | 15 | 15 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-Tracer FDG (F18 Fluorodeoxyglucose) PET/CT + Single-Tracer Cu64-DOTATATE PET/CT Exams | Single-Tracer FDG PET/CT + Single-Tracer Ga68-DOTATATE PET/CT Exams | Single-Tracer FDG PET/CT + Single-Tracer PSMA (Prostate-specific Membrane Antigen) PET/CT Exams | Total
Number analyzed (Participants) | 15 | 15 | 20 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.74 (19.74) | 54.25 (12.06) | 68.22 (11.74) | 60.84 (15.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 0 | 20
  Male | 3 | 7 | 20 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 14 | 17 | 46
  Unknown or Not Reported | 0 | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 15 | 13 | 16 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 20 | 50

OUTCOME MEASURES:

1. Primary Outcome: Completion of Two PET/CT Scans Per Patient as Dictated by Assigned Arm
Description: To obtain PET/CT imaging data suitable for developing new simultaneous dual-tracer PET techniques and processing algorithms for dual-tracer imaging of Fluorine-18 fluorodeoxyglucose (FDG) + Cu64-dodecane tetraacetic acid (DOTA) tyrosine-3-octreotate (TATE) (DOTATATE), FDG + Ga68-DOTATATE, and FDG + Ga68-prostate-specific membrane antigen (PSMA)-11 PET/CT
Time Frame: PET/CT exams were obtained on two separate days within a two week span.
Population: All participants enrolled on trial completed two different PET/CT scans within a two week span.
Measure: Count of Units; unit: PET/CT scans
Units Other Than Participants: PET/CT scans
Arm/Group | Single-Tracer FDG (F18 Fluorodeoxyglucose) PET/CT + Single-Tracer Cu64-DOTATATE PET/CT Exams | Single-Tracer FDG PET/CT + Single-Tracer Ga68-DOTATATE PET/CT Exams | Single-Tracer FDG PET/CT + Single-Tracer PSMA (Prostate-specific Membrane Antigen) PET/CT Exams
Number analyzed (Participants) | 15 | 15 | 20
Number analyzed (PET/CT scans) | 30 | 30 | 40
PET/CT scans | 30 | 30 | 40

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Single-Tracer FDG (F18 Fluorodeoxyglucose) PET/CT + Single-Tracer Cu64-DOTATATE PET/CT Exams | Single-Tracer FDG PET/CT + Single-Tracer Ga68-DOTATATE PET/CT Exams | Single-Tracer FDG PET/CT + Single-Tracer PSMA (Prostate-specific Membrane Antigen) PET/CT Exams
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/20
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT05680675/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT05680675/ICF_001.pdf